CLINICAL TRIAL: NCT05610735
Title: Combination Therapy With Liposomal Doxorubicin and Withaferin A (Ashwagandha, ASWD) in Recurrent Ovarian Cancer
Brief Title: Combination Therapy for Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sham Sunder Kakar (Other)
Collaborators: University of Louisville Health Care (Unknown)
Responsible Party: Sponsor-Investigator, Sham Sunder Kakar, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.0392
Record Dates: First submitted 2022-09-26; First posted 2022-11-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Ovarian Cancer
Keywords: DOXIL; Withaferin A; Ashwagandha; Recurrent Ovarian Cancer; Combination therapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; withaferin A; Ashwagandha

STUDY DESIGN:
Intervention Model Description: Recurrent Ovarian Cancer Participants treated with combination of DOXIL and Ashwagandha
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination of DOXIL and Ashwagandha (Experimental): The study contains two parts. In part 1 (Phase I), 18 patients with recurrent ovarian cancer will be recruited and administered IV with liposomal doxorubicin (DOXIL) 40 mg/m2 on day 1 of 28 days cycle for 4 cycles. Ashwagandha will be administered on daily basis for 2 years. Three doses of Ashwagandha (2 g, 4 g or 8.0 g) will be administered orally with water every day for two years to evaluate a tolerable dose of Ashwagandha. Six patients will be recruited for each dose.
  In part 2 Phase II), 54 additional patients with recurrent ovarian cancer will be recruited and administered with DOXIL IV (40 mg/m2) and maximum tolerable dose of Ashwagandha (determined from part 1) in the form tables orally with water on daily basis for two years. The survival rate (SR), complete response (CR) and partial response (PR) will be evaluated.
  Interventions: Drug: DOXIL; Drug: Withaferin A; Drug: Ashwagandha; Drug: Combination of ASWD and DOXIL

INTERVENTIONS:
Drug: DOXIL — DOXIL will be administered IV as 40 mg/m2 IV every four weeks for 4 cycles or until disease progression and/or unacceptable toxicity, whichever comes first to a maximum of 10 cycles.
  Other Names: Liposomal doxorubicin
Drug: Withaferin A — Ashwagandha in the form of tablets will be administered orally on daily basis.
  Other Names: Ashwagandha
Drug: Ashwagandha — Administered orally on daily basis twice a day
  Other Names: ASWD
Drug: Combination of ASWD and DOXIL — DOXIL administered IV once every four weeks. ASWD administered orally on daily basis, twice a day.
  Other Names: ASWD and DOXIL

SUMMARY:
The proposed study "combination therapy with liposomal doxorubicin and withaferin A (Ashwagandha, ASWD) in recurrent ovarian cancer" is focused to determine the feasibility and maximum tolerance dose of Ashwagandha with liposomal doxorubicin (DOXIL) in recurrent ovarian cancer patients. The study contains two parts. In part 1 (phase I), 18 patients with recurrent ovarian cancer eligible for DOXIL therapy will be recruited and three doses of Ashwagandha (2.0 g, 4.0 g and 8.0 g) in the form of tablets along with DOXIL will be evaluated for feasibility and tolerance of ASWD. In part 2 (phase II), 54 patients with recurrent ovarian cancer will be recruited and treated with DOXIL and Ashwagandha (dose determined from part 1) to evaluate the complete response (CR), partial response (PR), and stable disease (SD).

DETAILED DESCRIPTION:
Study Design Overview:

This is a two-part open-label clinical trial of ASWD (Ashwagandha) administered to patients with recurrent ovarian cancer in combination with liposomal doxorubicin, (DOXIL) following at least one previous line of chemotherapy. Patients will initially be enrolled in part 1 of the study, which is the feasibility/tolerability evaluation. Once the part 1 enrollment is completed, the patients will be enrolled in part 2 of the study.

In both parts, ASWD will be administered orally daily whereas liposomal doxorubicin will be administered intravenously (IV) every 4 weeks for at least 4 cycles or until disease progression and/or unacceptable toxicity, whichever comes first. If disease progression and/or unacceptable toxicity is not encountered, study treatment will be for a maximum of 10 cycles, or until a total cumulative dose of anthracycline therapy exceeds 450 mg/m2. Continued treatment with liposomal doxorubicin and/or ASWD will be determined by the provider. Once there is a completion of 10 cycles, ASWD will be continued in a daily regimen as maintenance, without continued liposomal doxorubicin, until disease progression and/or unacceptable toxicity.

Part 1 Part 1 (Phase I) is a feasibility/tolerability evaluation in which approximately 18 patients with recurrent ovarian cancer will be enrolled. The enrolled patients will be treated with 3 doses of ASWD [1.0 g, 2.0 g or 4.0 g/twice daily (total 2.0 g, 4.0 g or 8.0 g/day) taken orally with water in the form of capsule (500 mg/capsule, containing 500 mg of active ashwagandha)] in combination with set dosage of DOXIL (40 mg/m2 over 60 min, every 4 weeks). DOXIL will be administered at an initial rate of 1 mg/min to minimize the risk of infusion reactions. If no infusion related reactions occur, infusion rate will be increased to complete administration over 1 hour. Bolus injection or undiluted solution will not be administered.

Dose Escalation:

Approximately 18 subjects will be enrolled to escalating dose levels of ASWD in combination with DOXIL the approved dose of 40 mg/m2. Each dose level will initially enroll at least 3 DLT-evaluable subjects to a maximum of 6 subjects. Subsequent subjects, if any, assigned to receive the same dose level will be enrolled in groups of at least 2 DLT-evaluable subjects. Table 1 provides the dose escalation decision with target toxicity rate of 28.5% and optimal interval of (25.6%, 32.7%).

The ASWD starting dose level is 2.0 g, administered daily orally, starting with Cycle 1. The DOXIL dose level is fixed dose of 40 mg/m2 IV for every 4 weeks. The escalation dose of ASWD will be 4.0 g/day or 8.0 g/day for second and third cohort respectively and fixed dose of DOXIL. ASWD will be given alone if patient is no longer receiving DOXIL treatments. However, it will be given along with DOXIL if the patient continues DOXIL after 4 cycles.

The DLT observation period consists of the lead-in period [7 days of ashwagandha and Cycle 1 (21 days)] for 28 days total. To be considered DLT evaluate, subjects must complete at least 75% of ASWD dosing (i.e., at least 21 days) in the lead-in period and Cycle 1 or experience a DLT. DLT non-evaluate subjects may be replaced if needed to achieve the required number of DLT-evaluable subjects for dose escalation decisions. Dose-limiting toxicities will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (CTCAE v5.0). https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/ctcae_v5_quick_reference_5x7.pdf.

Ashwagandha is sold as an over-the-counter dietary supplement rich in WFA in 500 mg tablets containing 500 mg of active ashwagandha. ASWD will be provided by Marudhar Impex, Ahmedabad, India. Ashwagandha is manufactured and packed to capsules by Marudhar Impex under cGMP and analyzed by Eurofins Analytical Services India Private Limited. ASWD is extracted from the plant Withania somnifera grown under control conditions and packed in a Good Manufacturing Practices (GMPs) facility. It contains 0.71 % (w/w) Withanoside IV, 01.14% Withaferin A, 0.27% Withanoside V, 0.33% Withanone, 0.09% withanolide A, and 0.00% withanolide B determined by HPLC. The investigators will confirm the content of withaferin A using HPLC.

DOXIL is a liposomal formulation of doxorubicin hydrochloride encapsulated in liposomes with surface-bound methoxypolyethylene glycol (MPEG). Each liposomal doxorubicin vial contains pegylated liposomal doxorubicin HCl, 2 mg/mL and delivered as 10 ml (20 mg) in a concentrate for single dose intravenous infusion and is presented as sterile, translucent, and red suspension. For < 90 mg/m2, DOXIL is diluted in 250 ml Dextrose 5% in water and for > 90 mg/m2 DOXIL is diluted in 500 mL Dextrose in 5% in water. Aseptic technique must be strictly observed since no preservative or bacteriostatic agent is present in DOXIL. Diluted DOXIL should be refrigerated at 2°C to 8°C (36°F to 46°F) and administered within 24 hours.

Part 1 (Phase I) Part 1 of the study will be conducted using '3 + 3' traditional dose escalation design. Toxicities will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (CTCAE v5.0). Initially, 3 patients will be treated with 1.0 gram of ASWD twice daily (total of 2.0 grams/day) in combination with DOXIL, if none of them develop toxicity, then next 3 patients will be treated with 2.0 grams twice (total 4.0 grams/day) in combination with DOXIL, if none of them develop toxicity or has any issue, then next 3 patients will be treated with 4.0 grams twice daily (total 8.0 grams/day) in combination with DOXIL. If any of the patients has a Grade 3-4 hematologic or non-hematologic toxicity, the cohort will be expanded by three subjects (with a maximum of 6 patients at a given dose), prior to proceeding to the next dose. DOXIL dose will be 40 mg/m2 administered IV over a period of 60 min every 4 weeks for 4 cycles or until disease progression and/or unacceptable toxicity, whichever comes first to a maximum of 10 cycles. The total anthracycline (doxorubicin) cumulative dose should not exceed over 450 mg/m2.

AWSD will be administered on days 1-28 of each cycle. Patients will start ASWD on cycle 1, day 1 of DOXIL infusion. ASWD administration instructions will be provided to participants as follows:

"Take (appropriate number of capsules per dose escalation) tablets every 12 hours; to be initiated the day of starting chemotherapy." The medication may be taken with or without water and with or without food. If a dose is missed, it will not be re-taken. Participants will be instructed to keep a dose log. AWSD may be stored at ambient temperature protected from light at the participants' home. Plasma and urine samples will be collected for analysis of selected circulating biomarkers (proteins).

Part 2 (Phase II) Part 2 is an open label, exploration study to estimate the overall survival and response rate for participants treated daily with ASWD in the form of tablets in combination with DOXIL (40 mg/m2 IV for every 4 weeks for 4 cycles). Approximately 54 patients (including part 1 subjects treated with the highest feasible dose) will be enrolled in part 2 of the study. The enrollment for part 2 of the study will begin with the ASWD and liposomal doxorubicin dosages determined from part 1, provided no more than 2 out of 6 patients develop treatment related non-hematological toxicity in part 1 of the study. The enrolled patients will start taking ASWD capsules identified in part 1 for evaluation in part 2. Patients who participated in part 1 of the study will be offered to continue treatment to part 2, with a maximum tolerable dose. DOXIL will be administered every 4 weeks (40 mg/m2) for up to 10 cycles (limited to the standard limit of anthracycline administration, 450 mg/m2 cumulative dose of doxorubicin HCL). In the event of no progression and tolerance of the drug, patients should continue ASWD even DOXIL is stopped.

Dose Limiting Toxicities (DLT) The dose limiting toxicity window will include the first cycle of therapy (four weeks) and will be monitored prior to the initiation of cycle 2.

Laboratory values will be measured weekly during cycle one of therapy, then prior to each administration of DOXIL. These will include complete blood count (CBC) with platelets and complete metabolic panel (CMP) with liver function tests. In addition, prothrombin time and partial thromboplastin time will be monitored, simultaneously.

Hepatic Toxicity: Grade 3-4 hepatic toxicity will be defined as AST or ALT >3X upper limits of normal (ULN) and a concurrent bilirubin >2X ULN of any duration without finding of cholestasis (elevated alkaline phosphatase).

Hematologic Toxicity: Hematologic toxicity will be defined as: 1) Grade 4 neutropenia or thrombocytopenia > 7 days; 2) Grade 3 thrombocytopenia with bleeding; and 3) neutropenia fever.

Non-Hematologic Toxicity: Non-Hematologic toxicity will be defined as 1) Grade 4 alopecia, drug-related fever, and toxicities secondary to neutropenia and sepsis [with the exception of nausea and vomiting (if manageable with supportive care measures)], platelet count (< 25,000/mm3) 50 days beyond the start of the chemotherapy (not related to recurrent leukemia); 2) Grade 3 neurologic toxicity (sensory or autonomic).

Grade 3-4 non-hematologic toxicities will be considered a DLT and can be exempted from DLT if they resolve within 1 week, if they do not lead to hospitalization, and if they can be adequately managed with supportive care or conventional interventions within 72 hours.

Death: Any death not clearly due to underlying disease or extraneous causes

ELIGIBILITY:
Inclusion Criteria:

Patients with recurrent ovarian/fallopian tube/primary peritoneal cancer for whom liposomal Doxorubicin would be an acceptable therapeutic option will be recruited. Patients are eligible if they have received first line chemotherapy containing platinum and have become platinum resistance or have refractory disease. The patient must also meet all the following criteria:

1. Signed approved informed consent document stating that they understand the investigational nature of the treatment program before entering study
2. Female patients, age ≥ 18 years
3. Pathological confirmed ovarian, fallopian tube, or primary peritoneal carcinoma with the one of the following histologic types: high grade papillary serous carcinoma, low grade papillary serous carcinoma, high grade mucinous carcinoma, low grade mucinous carcinoma, clear cell carcinoma, high grade endometrioid carcinoma.
4. Received at least one line chemotherapy, which must be a platinum containing regimen and develop platinum resistance. Patients may have not received previous liposomal doxorubicin therapy, and must be considered to be eligible for single agent liposomal doxorubicin treatment.
5. Patients may have undergone surgical cytoreduction at the time of primary diagnosis or following neoadjuvant chemotherapy. Patients who had optimal (<1 cm residual disease) or suboptimal (>1 cm residual disease) following surgical cytoreduction will be included.

   Patients who did not undergo surgical cytoreduction will also be included.
6. Recurrent disease confirmed by biopsy, radiologic imaging, and/or elevated CA 125
7. Patients may have received radiation therapy
8. Life expectancy > 6 months
9. Part 1: Have evaluable disease by radiologic measurements (See 11) or CA 125
10. Part 2: Have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as > 1 cm on cross-sectional imaging (where the CT slice thickness is no greater than 5 mm) or at least 2 cm by standard techniques; positron emissions tomography (PET] and ultrasound are not permitted methods for tumor measurements under this protocol. Consult RECIST 1.1 guidance for additional information (Appendix C and Eisenhauer et al., 2009; Ref 61).
11. Adequate organ function within 14 days prior to first WFA/ASWD dose or liposomal doxorubicin whichever occurs first, including the following: absolute neutrophil count (ANC) ≥ 1.5 x 103/L, platelet count ≥ 100 x 103/L, hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L), patients may receive packed RBC transfusion to achieve this level at the discretion of the investigator, total bilirubin < 1.5 x upper limit of normal (ULN) unless elevated secondary to conditions such as Gilbert's Disease, aspartate aminotransferase (AST) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases), alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases), alkaline phosphatase < 3.0 x ULN, calculated creatinine clearance ≥ 60 mL/min per Cockcroft and Gault formula
12. Satisfy one of the following:

    * Females: non-pregnant and non-lactating; surgically sterile, post- menopausal, or patient/partner compliant with a reliable contraceptive regimen, as determined by the investigator, for 4 weeks prior to screening.
    * Patients of reproductive potential must test negative for pregnancy at screening, prior to each cycle, and must agree to use a reliable method of birth control during the study period and 6 months following completion of treatment.
13. The patient is willing and able to comply with the study visit schedule and procedures and has geographical proximity (Investigator's discretion) that allows follow-up specified by the protocol
14. For Part 1: Patients have discontinued all prior chemotherapies, biological therapies, and other investigational therapies for cancer for at least 4 weeks prior to study treatment and have recovered from the acute effects of therapy
15. ECOG performance status of 0, 1, or 2
16. Adequate ejection fraction determined by transthoracic echo or MUGA of at least 55%
17. Patients may have received prior anthracycline or anthracenedione therapy. In this scenario, the use of prior treatments will be incorporated into the cumulative dose calculations when applicable, given a known increased risk of cardiomyopathy to 11% when the cumulative dose of liposomal doxorubicin was between 450 mg/m2 to 550 mg/m2.

    -

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. ECOG performance status 3 or 4
2. Pregnant or breastfeeding
3. Treatment with another investigational drug, biological agent, or device within 4 weeks (6 weeks for biological agents) before screening or 5 half-lives of study agent, whichever is longer
4. Patients with treated or untreated parenchymal brain metastases or leptomeningeal disease. Brain imaging is required for symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients
5. Patients with known pericardial effusion
6. Patients with active infection or serious concomitant systemic disorder (for example, heart failure) incompatible with the study (at the discretion of the Investigator)
7. Presence or history of malignancy other than ovarian cancer that does not include carcinoma in situ of the cervix, or non-melanoma skin cancer. In the case of other malignancies, patients may be considered for participation if the prior malignancies were diagnosed and definitively treated at least two years previously with no subsequent evidence of recurrence
8. Presence of an underlying disease state associated with active bleeding
9. Concurrent treatment with other anticancer drugs
10. Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device
11. Patients with any other medical conditions that, in the opinion of the Investigator, would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
12. Patients with known septicemia, severe infection, or acute hepatitis
13. Patients with known congestive heart failure or unstable angina or those who had a myocardial infarction within the past 6 months
14. Patients with known clinically significant pericardial disease
15. Patients taking medications known to affect the cardiac conduction system
16. Allergy to WFA/ASWD
17. Previous treatment with liposomal doxorubicin
18. Prior use of other anthracyclines or anthracenediones -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pathological confirmed ovarian, fallopian tube, or primary peritoneal carcinoma with the one of the following histologic types: high grade papillary serous carcinoma, low grade papillary serous carcinoma, high grade mucinous carcinoma, low grade mucinous carcinoma, clear cell carcinoma, high grade endometrioid carcinoma, undifferentiated carcinoma, mixed epithelial carcinoma, and adenocarcinomas not otherwise specified
Enrollment: 72 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From study entry to time of progression or death, whichever occurs first, assessed up to 4 years.
  Will be presented by Kaplan Meier methods.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | From study entry, up to 4 years.
  All adverse events, including severe adverse events and treatment-related adverse events, will be categorized and graded for severity according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Objective response rate (ORR) | From the start of the treatment until disease progression/recurrence, assessed up to 4 years
  Quantified as the binomial proportion of patients with measurable disease at enrollment who have a best overall response of complete response (CR) or partial response (PR).
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 4 years.
  Will be defined among participants with the best overall response of complete response (CR) or partial response (PR). Will be presented by Kaplan Meier methods.
Overall survival | Time from study entry to date of death from any cause, assessed up to 4 years
  Will be presented by Kaplan Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Goldsberry, MD, Principal Investigator — Brown Cancer Center at University of Louisville
Locations (1):
- UofL Health Brown Cancer Center, Louisville, Kentucky, United States